CLINICAL TRIAL: NCT03993418
Title: Physiological Effects of Long-term Consumption of Non-nutritive Sweeteners in Humans: a Pilot 12 Week Randomised Trial
Brief Title: Physiological Effects of Stevia Consumption in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Lancaster University (Other)
Responsible Party: Principal Investigator, Nikoleta Stamataki, PhD student, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 4812
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Glucose Intolerance; Obesity
MeSH Terms: conditions — Glucose Intolerance; Obesity | interventions — stevioside

STUDY DESIGN:
Intervention Model Description: 2-group parallel 12-week intervention study with control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stevia arm (Experimental): stevia drops
  Interventions: Dietary Supplement: stevia
- Control arm (No Intervention): No change in diet

INTERVENTIONS:
Dietary Supplement: stevia — This arm will be required to consume 5 stevia drops twice daily in habitual drinks
  Arms: Stevia arm

SUMMARY:
This study will evaluate whether long-term consumption of the low calorie sweetener stevia affects glucose tolerance in healthy participants. With regard to this aim, we will recruit 2 study groups, the stevia group where participants will be required to add stevia drops twice daily in their habitual drinks and the control group where participants will be asked not to change anything in their diet and lifestyle.

DETAILED DESCRIPTION:
Excess consumption of caloric sweeteners contributes to the alarming rates of overweight and obesity, whereas non-nutritive sweeteners (NNS) are non-caloric alternatives offering sensory and health benefits. NNS are widely used to moderate energy intake and postprandial glycaemia, but there is controversial evidence about their role and effects. Stevia, a natural NNS, has been suggested to assist with glucose regulation but data on glucose tolerance after daily consumption of stevia are lacking. The investigators plan to undertake a pilot randomized 2-parallel arm open-label 12-week trial, where participants will start consuming stevia with their habitual drinks. Thirty healthy volunteers (not habitual consumers of stevia or other NNS) will be recruited. The intervention group (n=15) will consume 5 drops of stevia with their habitual drinks twice daily whereas the control group (n=15) will not be required to change anything in their diet, but avoid consuming NNS or diet beverages for the study duration.

Key measures in glucose homeostasis including glucose response to an oral glucose tolerance test will be performed before and after the intervention period. Serum and plasma samples will be stored for potential analysis of insulin and gut hormones levels.

Participants will have to attend 3 study visits, visit week 0, visit week 6 and visit week 12, but the primary outcome will be assessed in visit week 0 and visit week 12.

Participants will be weighed; dietary intake, physical activity and appetite will be also assessed. Faecal samples will be collected and gut microbiome analysis may be performed. Gut microbiome has been considered to be a key linked topic, since it has been suggested that saccharin consumption may induce glucose intolerance in humans through alterations in gut microbiota in humans.

The trial will assess whether regular use of stevia in realistic amounts has any effects on glucose homeostasis, and aims to elucidate our understanding of long-term physiological effects of NNS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* BMI 18.5-25 kg/m2
* No or low NNS consumers (up to 1 can of diet soda per week or 1 sachet of NNS per week)
* DEBQ for restraint eating ≤ 3
* Healthy - general good health
* Not taking medications that affect metabolism or appetite (i.e. thiazide diuretics, glucocorticoids or beta blockers)
* Stable weight, ≤ 5 kg last 12 months
* Fasting blood glucose ≤6.0 mmol/L
* Willing to comply with the study protocol
* No self-reported food allergy or intolerance to foods supplied during the study
* The participant is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* The participant is able to read, comprehend and record information written in English.
* A signed and dated written informed consent is obtained from the participant.

Exclusion Criteria:

* Age under 18 years or over 40 years old.
* BMI >25 kg/m2 and <18.5kg/m2
* Participants who are not willing to comply with study procedures (including expression of dislike for NNS)
* Habitual NNS consumers, >1 can of diet beverage or >1 sachet of low calorie sweeteners per week.
* Fasting blood glucose measured > 6 mmol/L
* Subjects who are currently dieting and having ceased a diet in < 4 weeks
* DEBQ score for restraint eating > 3
* Subjects who follow special diets for weight maintenance, such as Atkins Diet, Weight Watchers, gluten-free diet, The Zone diet, Vegetarian Diet, Raw Food Diet etc.
* Vegetarians, vegans
* Subjects who take recreational substances such as cannabis.
* Presence of any chronic condition requiring medication that might affect our results (e.g. diabetes, mental diseases, gastrointestinal diseases)
* Subjects with eating disorders (binge eating disorder, bulimia etc)
* Subjects who are currently experiencing anxiety or depression
* Participants who drink alcohol more than the NHS guidelines (14 units per week)
* >10 h of vigorous physical activities per week and/or planning to increase/decrease physical activity levels in the next months.
* Having ceased smoking in the last six months
* Female participants who are, or may be, pregnant, or currently lactating.
* Subjects who regularly consume dietary supplements for weight loss, muscle building etc.
* Subjects with food allergies or intolerances related to the study.
* Subjects who have given blood elsewhere within the last month.
* The participant cannot read, comprehend and record information written in English.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Glucose response to an oral glucose tolerance test (OGTT) measured as incremental area under the curve (iAUC) | Week 0 and week 12
  blood glucose levels will be measured at baseline (0) and at 15, 30, 45, 60, 90 and 120 min after the consumption of a 75 g glucose load and iAUC will be calculated

SECONDARY OUTCOMES:
Change in body weight | Week 0, visit week 6 and week 12
  body weight will be measured on visit week 0, visit week 6 and visit week 12
Change in dietary intake | Week 0, visit week 6 and week 12
  participants will fill out 3 days of diet recalls before coming to all 3 study visits using Intake24
Change in waist circumference | Week 0, visit week 6 and week 12
  waist circumference will be measured on visit week 0, visit week 6 and visit week 12
Change in appetite | Week 0 and week 12
  Appetite questionnaires (three factor eating questionnaire, sweet food frequency questionnaire, Satiety, hunger, and food cravings - using the Control of Eating Questionnaire ) will be completed on visit week 0 and visit week 12
Change in fasting blood glucose | Week 0 and week 12
  Fasting blood glucose will be measured on visit week 0 and visit week 12.
Change in the 75-OGTT 2-hour blood glucose | Week 0 and week 12
  75g OGTT 2-h blood glucose will be measured on visit week 0 and visit week 12.

OTHER OUTCOMES:
Physical activity | Week 0, visit week 6 and week 12
  Total MET-minutes per week measured via the International Physical Activity Questionnaire (IPAQ).
Physical activity | Week 0, week 6, week 12
  Number of steps per day. 3 days before visit week 0, visit week 6 and visit week 12
Blood pressure | Week 0, visit week 6 and week 12
  Blood pressure will be measure on visit week 0, visit week 6 and visit week 12
Composition of gut microbiome | Week 0 and week 12
  Changes in gut microbiota will be measured by 16S rRNA gene sequencing. This outcome is optional and will be decided by the investigators based on the findings in the primary outcome.
Fasting plasma insulin | Week 0 and week 12
  This outcome is optional and will be decided by the investigators based on the findings in the primary outcome
75g OGTT derived iAUC plasma insulin | Week 0 and week 12
  This outcome is optional and will be decided by the investigators based on the findings in the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: John McLaughlin, Principal Investigator — University of Manchester
Locations (1):
- University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided